CLINICAL TRIAL: NCT06919497
Title: NOICE vs. Nothing | Thermode: A Prospective, Randomized, Crossover Study
Brief Title: NOICE vs. Nothing | Thermode
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 80078
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Spatial Audio Stimulation
Keywords: Thermal Sensory Analyzer (TSA-II); Peltier-Based Contact Thermode

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spatial audio stimulation (Experimental): Participant will receive spatial audio stimulation first and then will not receive spatial audio stimulation in the latter part of the study.
  Interventions: Behavioral: Spatial audio stimulation; Behavioral: No spatial audio stimulation
- No spatial audio stimulation (Experimental): Participant will not receive spatial audio stimulation first and then will receive spatial audio stimulation in the latter part of the study.
  Interventions: Behavioral: Spatial audio stimulation; Behavioral: No spatial audio stimulation

INTERVENTIONS:
Behavioral: Spatial audio stimulation — Study RA will affix the thermode to the dorsum of the participant's dominant or non-dominant hand. Participants will undergo heat-pain-inducing thermode exposure. The intervention will be randomized to receive spatial audio stimulation or not for the first HPT trial, then crossed over to the other study condition for the second HPT trial.
  Participants will be randomized to expose their dominant or non-dominant hand first. Between each levels test, the thermode will be moved to the other hand (ex: VR: DH, NDH, DH; Nothing: NDH, DH, NDH). There will be a 30 second break between each levels test and a five-minute washout period between each intervention.
Behavioral: No spatial audio stimulation — Study RA will affix the thermode to the dorsum of the participant's dominant or non-dominant hand. Participants will undergo heat-pain-inducing thermode exposure. The intervention will be randomized to receive spatial audio stimulation or not for the first HPT trial, then crossed over to the other study condition for the second HPT trial.
  Participants will be randomized to expose their dominant or non-dominant hand first. Between each levels test, the thermode will be moved to the other hand (ex: VR: DH, NDH, DH; Nothing: NDH, DH, NDH). There will be a 30 second break between each levels test and a five-minute washout period between each intervention.

SUMMARY:
The purpose of this study is to test whether the non-visual immersive technologies, which uses spatial audio simulation, can help people better tolerate heat pain. As a proof-of-concept study, study team will use the NOICE device. This research is not studying the NOICE device specifically and the device is not a medical device.

DETAILED DESCRIPTION:
This study addresses the research gap in understanding how spatial audio impacts pain perception, specifically heat pain, in clinical settings. It is important to explore this because spatial audio may serve as a non-pharmaceutical, immersive alternative to traditional visual-based distraction methods like virtual reality.

The investigators hypothesize that participants using the spatial audio simulation device will report an increased heat pain threshold compared to not using the device. This knowledge could improve information on the perception of pain for participant who prefer not to use VR headsets.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years and older
* English-speaking
* Intact hearing
* No self-reported or clinically diagnosed acute or chronic medical conditions that affect safe participation

Exclusion Criteria:

* Use chronotropic heart medications
* Use pain medications
* Current hearing loss
* Currently taking beta blockers, or opioids or other prescription pain medications
* History of chronic pain or acute pain syndromes
* Current hearing loss

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in heat pain threshold | Duration of intervention, approximately 15 minutes
  Heat pain threshold measured by the TSA Air II device. Temperature ranges from 32 degrees C to 44 degrees C, with higher temperatures indicating a higher heat pain threshold.

SECONDARY OUTCOMES:
Change in heat pain sensitivity (HPS) | immediately after intervention
  To evaluate heat pain sensitivity(HPS), participants will complete the Numerical Rating Pain Scale (NRPS) immediately following each trial, where they rank pain sensitivity on an ordinal scale from 0 = no pain to 10 = worst pain possible under both treatment conditions.
Anxiety Level | immediately after intervention
  participants will complete the Visual Analog Scale for Measuring Anxiety (VAS-A) immediately following each group of levels tests, where they will rank anxiety scores on a sliding scale from 0 = No anxiety/fear to 100 = Worst possible anxiety/fear
ISO Ergonomic scale | immediately after intervention
  The scale has 6 items. Scores ranges from 1-5 (1 = strongly disagree and 5 = strongly agree)
System Usability Scale (SUS) Score | immediately after intervention
  The scale has 10 items. Scores ranges from 1-5 (1 = strongly disagree and 5 = strongly agree)
Device satisfaction | immediately after intervention
  To evaluate the overall impact of device satisfaction of the spatial audio stimulation device, participants will complete the Patient Technology Satisfaction Survey. Participants will rank each factor on a Likert scale from 1 = not at all to 5 = completely.

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States